CLINICAL TRIAL: NCT02714790
Title: Ruolo Prognostico Della Malattia Minima Residua Nella Leucemia Mieloide Acuta
Brief Title: Prognostic Role of Minimal Residual Disease in Acute Myeloid Leukemia
Acronym: LAM-MMR
Status: Completed | Type: Observational
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Ernesta Audisio, MD, A.O.U. Città della Salute e della Scienza
Other Study IDs: LAM-MMR
Record Dates: First submitted 2016-03-03; First posted 2016-03-22 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Acute Myeloid Leukemia; Minimal Residual Disease; Wilms Tumor
Keywords: Acute Myeloid Leukemia; Minimal Residual Disease; Wilms Tumor
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm, Residual; Wilms Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Study purpose is to assess the prognostic role of Minimal Residual Disease (defined as medullary expression of WT1 gene), performed at Baseline and during treatment according to clinical practice. MRD results will be relate to treatment outcome and survival analysis variables (Overall Survival, Disease Free Survival, Cumulative Incidence of Relapse)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Acute Myeloid Leukemia
* Age > 18 years
* Intensive chemotherapy as first line curative treatment
* Observation period: March 2004 - September 2014
* Bone marrow WT1 expression and Immunophenotyping by multi-parametric flow cytometry performed at baseline
* Written informed consent

Exclusion Criteria:

* Diagnosis of Acute Promyelocytic Leukemia
* Bone marrow WT1 expression and Immunophenotyping by multi-parametric flow cytometry NOT performed at baseline
* Patient ineligible to intensive chemotherapy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with new diagnosis of acute myeloid leukemia treated with intensive chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2015-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Response | +28 days after End of induction chemotherapy - Before Allogeneic Transplant, average of 3 to 6 months from beginning of therapy
  Complete remission after chemotherapy

SECONDARY OUTCOMES:
Disease Free Survival | +28 days after End of induction chemotherapy -Before Allogeneic Transplant, average of 3 to 6 months from beginning of therapy - +30 days after Allogeneic Transplant - Date of Relapse for at least 1 year (up to 10 years)
  Date of relapse or date of remission status
Overall Survival | Date of last follow-up for at least 1 year (up to 10 years) or Death
  Time to last follow-up or death
Cumulative Incidence of Relapse | Date of Allogeneic Transplant, Date of Relapse for at least 1 year (up to 10 years - assessed every 3 months), Date of last follow-up for at least 1 year (up to 10 years) or Death
  CIR was calculated from the date of allo-HCT to the date of relapse or the date of the last follow-up, with death without relapse as a competing event.

CONTACTS AND LOCATIONS:
Overall Officials: Ernesta Audisio, MD, Principal Investigator — AO Città della Salute e della Scienza di Torino

IPD SHARING:
Plan to Share IPD: Yes
paper publication

REFERENCES:
- [Derived] Frairia C, Aydin S, Audisio E, Riera L, Aliberti S, Allione B, Busca A, D'Ardia S, Dellacasa CM, Demurtas A, Evangelista A, Ciccone G, Francia di Celle P, Nicolino B, Stacchini A, Marmont F, Vitolo U. Post-remissional and pre-transplant role of minimal residual disease detected by WT1 in acute myeloid leukemia: A retrospective cohort study. Leuk Res. 2017 Oct;61:10-17. doi: 10.1016/j.leukres.2017.08.008. Epub 2017 Aug 30. PMID 28846953